CLINICAL TRIAL: NCT02833064
Title: Identification of Outcome Biomarkers in Patients With Liver Failure.
Brief Title: Biomarkers in Liver Failure
Status: Active, not recruiting | Type: Observational
Sponsor: University of Edinburgh (Other)
Collaborators: NHS Lothian (Other Government)
Responsible Party: Sponsor
Other Study IDs: AC16086
Record Dates: First submitted 2016-07-11; First posted 2016-07-14 (Estimated); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Acute Liver Failure; Acute Liver Injury; Acute on Chronic Hepatic Failure
MeSH Terms: conditions — Liver Failure, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Acute Liver Failure: * biological sampling
  * MRI scanning for patients with paracetamol induced acute liver failure
  Interventions: Radiation: Non-contrast magnetic resonance imaging; Other: Biological sampling
- Acute Liver Injury: - biological sampling
  Interventions: Other: Biological sampling
- Acute on Chronic Hepatic Injury: - biological sampling
  Interventions: Other: Biological sampling
- Stable Cirrhotics: - biological sampling
  Interventions: Other: Biological sampling
- Non-cirrhotic liver disease: - biological sampling
  Interventions: Other: Biological sampling

INTERVENTIONS:
Radiation: Non-contrast magnetic resonance imaging
  Groups: Acute Liver Failure
Other: Biological sampling — Blood, urine, stool and breath sampling and analysis

SUMMARY:
Acute liver injury (ALI) and acute liver failure (ALF) are rare clinical conditions, the latter often associated with a poor outcome. To improve outcomes for these patients, clinicians need to develop a clearer understanding of the pathophysiology of this condition. Biomarkers and novel imaging techniques are vital to investigating and understanding the pathophysiology of ALI. Patients with ALI or ALF aged over 16 and due to any cause will be eligible to take part in the study. The study will involve collection of biological samples (blood, urine, stool and breath) from included patients once daily for up to 7 days. For patients undergoing liver transplantation, a small sample of explanted (removed) liver tissue will be obtained. A small subgroup of patients with paracetamol induced acute liver failure will be eligible to be included in a pilot MRI (magnetic resonance imaging) study, which will involve two MRI scans during the first 7 days of their admission. All patients will be recruited from the Royal Infirmary of Edinburgh.

DETAILED DESCRIPTION:
For inpatients, the investigators wish to collect biological samples from each patient once daily for the first seven days of their admission. 25mls of blood will be taken daily for research purposes, at the same time at routine clinical samples to reduce discomfort from additional venepuncture. One urine sample will be taken daily (which can be taken from a catheter if the patient has a catheter in place), and a sample of stool if the patient moves their bowels. The investigators wish to collect breath for analysis, at one point during the first seven days of admission. Breath analysis requires the patients to be fasted for four hours (with the exception of water) prior to the test. If the patient undergoes liver transplantation during their admission, a small sample of explanted liver tissue will be obtained for later analysis.

For outpatients (acute liver injury, stable cirrhotics, non-cirrhotic liver disease), the investigators will ask them to attend the ward or the outpatient department for collection of biological samples. The investigators will take 25 mls of blood as above, along with a urine and stool sample if they are able to provide this at their first attendance. Breath analysis will also be undertaken during this visit to the hospital, after a 4 hour fast (with the exception of water). Outpatients will then be asked to return one month later, when further blood (25mls), urine and stool samples will be collected.

As a pilot study, the investigators wish to perform MRI scanning on a subset of 10 patients with paracetamol induced acute liver failure. Paracetamol induced acute liver failure is associated with a particularly rapid course, characterised by hepatic encephalopathy and renal impairment. In view of the potential for renal impairment, intravenous contrast will not be used for these scans, but alternative techniques employed such as artertial spin labelling.

The participant does not need to consent to each individual part of the study to be able to take part.

ELIGIBILITY:
Inclusion Criteria:

* acute liver injury (newly deranged liver function tests (LFTs) and coagulopathy with International Normalized Ratio (INR) >1.5 in absence of chronic liver disease)
* acute liver failure ( as above, plus hepatic encephalopathy)
* acute on chronic liver failure (worsening of LFTS and development of at least 1 organ failure in patient with cirrhosis)
* stable cirrhosis
* non-cirrhotic liver disease

Exclusion Criteria:

* refusal of consent
* withdrawal of consent

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: 1. Acute liver failure
  2. Acute liver injury
  3. Acute on chronic hepatic failure
  4. Stable cirrhotics
  5. Non-cirrhotic liver disease
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-11-28 (Actual); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Identification of biomarkers and radiological markers predictive of development of complications and outcomes in acute liver injury and acute liver failure. | 10 years

SECONDARY OUTCOMES:
Identification of proteins involved in the pathogenesis of acute liver injury and acute liver failure | 10 years

IPD SHARING:
Plan to Share IPD: Undecided